CLINICAL TRIAL: NCT01698684
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of Avanafil for On-Demand Treatment of Men With Erectile Dysfunction
Brief Title: Research Evaluating a PDE5 Inhibitor for Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TA-501
Record Dates: First submitted 2012-09-25; First posted 2012-10-03 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Avanafil 100 mg (Experimental)
  Interventions: Drug: Avanafil 100 mg
- Avanafil 200 mg (Experimental)
  Interventions: Drug: Avanafil 200 mg

INTERVENTIONS:
Drug: Placebo — One dose 15 minutes before attempting intercourse
  Arms: Placebo
Drug: Avanafil 100 mg — One dose 15 minutes before attempting intercourse
  Arms: Avanafil 100 mg
Drug: Avanafil 200 mg — One dose 15 minutes before attempting intercourse
  Arms: Avanafil 200 mg

SUMMARY:
The objectives of this study are to examine the therapeutic effects of two doses of avanafil after dosing in men with erectile dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 18 years of age;
* Minimum 6 months of erectile dysfunction;
* In a monogamous, heterosexual relationship for at least 3 months;
* Agree to make at least 4 attempts at intercourse per month;
* Provide written informed consent;
* Agree not to use any other ED treatments for erectile dysfunction;
* Willing and able to comply with all study requirements.

Exclusion Criteria:

* Allergy or hypersensitivity to PDE5 inhibitors;
* History of dose-limiting AEs with a PDE5 inhibitor or discontinued use of a PDE5 inhibitor;
* Concomitant use of one or more of the following medications:

  * Other prescription or OTC drugs known to interfere with metabolism by the CYP 3A4 enzyme;
  * Dose of an alpha blocker that has not been stable for at least 14 days;
  * Any nitrate;
* ED as a consequence of advanced neurologic disease, spinal cord injury,or radical prostatectomy;
* Myocardial infarction, stroke, life-threatening arrhythmia or coronary revascularization within the past 6 months;
* Unstable angina, angina with sexual intercourse, or congestive heart failure > NYHA Class II;
* Poorly controlled type 1 or type 2 diabetes;
* Evidence of prostate cancer or previous radical prostatectomy;
* Untreated hypogonadism or total testosterone levels outside normal reference range;
* Abnormal laboratory value(s) judged to be clinically significant by the investigator;
* Positive urine drug screen;
* History of retinitis pigmentosa, nonarteritic anterior ischemic optic neuropathy or glaucoma;
* Previous participation in any other study with avanafil;
* Use of any other investigational medication or device for any indication within 30 days prior to enrollment or at any time during this study;
* Evidence of any clinically significant medical, psychiatric, social or other condition by history, physical examination or laboratory studies that, in the opinion of the investigator, would contraindicate the administration of study medications, affect compliance, interfere with study evaluations, limit study participation, contraindicate sexual activity or confound the interpretation of study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chuck Bowden, M.D., Study Director — VIVUS LLC
Locations (3):
- United States (3):
  - Jupiter, Florida
  - Raleigh, North Carolina
  - Wilmington, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Started | 145 | 147 | 148
ITT Population | 136 | 139 | 139
Safety Population | 143 | 146 | 146
Completed | 116 | 124 | 127
Not Completed | 29 | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg | Total
Number analyzed (Participants) | 145 | 147 | 148 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.92) | 58.5 (10.19) | 57.9 (10.61) | 58.2 (10.23)
Age, Customized [Number; unit: participants]
  <50 Years | 29 | 25 | 29 | 83
  >=50 to <65 Years | 74 | 78 | 76 | 228
  >=65 Years | 42 | 44 | 43 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 145 | 147 | 148 | 440
Race/Ethnicity, Customized [Number; unit: participants]
  White | 102 | 107 | 124 | 333
  Black or African American | 37 | 35 | 22 | 94
  Asian | 3 | 3 | 1 | 7
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Multiple Races | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 145 | 147 | 148 | 440

OUTCOME MEASURES:

1. Primary Outcome: Per-subject Proportion of Sexual Attempts That Had an Erectogenic Effect Within Approximately 15 Minutes Following Dosing
Time Frame: Week 0 (Baseline) up to Week 8 (End of Study)
Population: The intent-to-treat (ITT) population consists of all subjects who are randomized, take at least 1 dose of study medication, and have at least 1 post-dose efficacy assessment.
Measure: Mean (Standard Deviation); unit: percentage of successes
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 136 | 139 | 139
percentage of successes | 14.9 (25.1) | 25.9 (32.0) | 29.1 (34)

ADVERSE EVENTS:
Time Frame: Approximately 16 weeks (from written informed consent provided and until 28 calendar days after the last dose of the study drug was administered, or until the subject was discontinued from the study, whichever was later)
Description: The safety population includes all subjects who receive at least 1 dose of study medication and have any safety data available.
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Serious Adverse Events (participants affected / at risk) | 2/143 | 4/146 | 3/146
Other Adverse Events (participants affected / at risk) | 13/143 | 7/146 | 26/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=143) | Avanafil 100 mg (N=146) | Avanafil 200 mg (N=146)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=143) | Avanafil 100 mg (N=146) | Avanafil 200 mg (N=146)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 13 (37)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (9)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 3 (3) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days